CLINICAL TRIAL: NCT02072824
Title: A Double-blind, Placebo-controlled, Parallel-group, Multicenter Study Of The Efficacy And Safety Of Pregabalin As Adjunctive Therapy In Children 1 Month Through <4 Years Of Age With Partial Onset Seizures
Brief Title: A Safety, Efficacy, and Tolerability Trial of Pregabalin as Add-On Treatment in Pediatric Subjects <4 Years of Age With Partial Onset Seizures.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081042; 2013-003420-37 (EudraCT Number)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2018-09

CONDITIONS: Partial Onset Seizures
Keywords: Partial Onset Seizures; Epilepsy; Safety; Efficacy; Tolerability; Pregabalin; Lyrica; Adjunctive treatment; Placebo controlled; blinded; Eligibility Criteria
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study Drug Level 1 (Experimental)
  Interventions: Drug: Pregabalin Dose Level 1
- Study Drug Level 2 (Experimental)
  Interventions: Drug: Pregabalin Dose Level 2
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin Dose Level 1 — Pregabalin liquid dosed daily three times a day in equally divided doses escalated to 7.0 mg/kg/day beginning at Randomization through Taper Phase then tapered to 3.5 mg/kg/day during 1 week Taper Phase
  Arms: Study Drug Level 1
Drug: Pregabalin Dose Level 2 — Pregabalin liquid dosed daily three times a day in equally divided doses escalated to 14.0 mg/kg/day beginning at Randomization through Taper Phase then tapered to 3.5 mg/kg/day during 1 week Taper Phase
  Arms: Study Drug Level 2
Drug: Placebo — Placebo Liquid dosed three times daily beginning at Randomization through Taper Phase
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the effectiveness of 2 doses of pregabalin to reduce seizure frequency as an add on therapy in pediatric subjects 1 month to <4 years of age with refractory partial onset seizures. It is hypothesized that both doses of pregabalin will demonstrate superior efficacy when compared to placebo by reducing the partial onset seizure frequency and that pregabalin will be safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have 3 partial onset seizures in the month prior to screening.
* Subject must have 2 partial onset seizures during the 48 hour baseline phase.
* Signed Informed Consent.
* On 1-3 stable anti-epileptic drugs at screening.

Exclusion Criteria:

* Primary generalized seizures including clonic, tonic, clonic-tonic, absence, febrile seizures, and infantile spasms.
* Lennox-Gasteau, BECTS, and Dravet's syndrome.
* Status epliepticus within 1 year of screening.
* Any change in AED regimen with 7 days of screening.
* Progressive structural central nervous system (CNS) lesion or a progressive encephalopathy.
* Progressive errors of metabolism.

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (69):
- United States (5):
  - Pediatric Epilepsy Center of Central Florida, Orlando, Florida
  - Pediatric Neurology, PA, Orlando, Florida
  - Pediatric Epilepsy & Neurology Specialists, PA, Tampa, Florida
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
- GU Republican Scientific and Practical Center Mother and Child, Minsk, Belarus
- UZ Brussel, Brussels, Brussels Capital, Belgium
- University Clinical Centre of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Bulgaria (2):
  - UMHAT Dr. Georgi Stranski Ltd., Pleven
  - UMHAT "Sveti Georgi" Ltd., Plovdiv
- China (3):
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Beijing Children's Hospital, Beijing
- Hopital Raymond Poincare, Garches, France
- Universitaetsklinikum Jena, Jena, Thuringia, Germany
- Greece (2):
  - University General Hospital Attikon, Athens
  - General Hospital of Thessaloniki Ippokratio, Thessaloniki
- Hungary (6):
  - Dr. Kenessey Albert Korhaz es Rendelointezet, Balassagyarmat
  - Szent János Kórház es Észak Budai Egyesitett Kórházak, Budapest
  - Szent Margit Kórház, Budapest
  - Semmelweis Egyetem, I. Sz. Gyermekgyogyaszati Klinika, Budapest
  - Magyarorszagi Reformatus Egyhaz Bethesda Gyermekkorhaz, Gyermekneurologia, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
- Israel (4):
  - Pharmacy of The E. Wolfson Medical Center, Holon
  - The E. Wolfson Medical Center, Holon
  - Pharmacy of Tel Aviv Sourasky Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Lebanon (2):
  - American University of Beirut Medical Center, Beirut
  - Saint George Hospital - University Medical Center, Beirut
- Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan, Malaysia
- Philippines (7):
  - Cebu Doctors' University Hospital, Cebu City, CEBU
  - Perpetual Succour Hospital, Cebu City, CEBU
  - Manila Doctors Hospital, Manila
  - Metropolitan Medical Center, Manila
  - University of Santo Tomas Hospital, Manila
  - St. Luke's Medical Center, Quezon City
  - Philippine Children's Medical Center, Quezon City
- Romania (2):
  - Centrul Medical Unirea, Bucharest
  - Spitalul Clinic de Urgente pentru Copii "Sf. Maria", Iași
- Russia (11):
  - Nizhmedklinika, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Perm State Medical University n. a. acad. E.A. Vagner, Perm, Permskiy KRAY
  - FSFEI HE N.I. Pirogov RNRMU of Minzdrav of Russia, Moscow
  - Perm State Medical University n. a. acad. E.A. Vagner, Perm
  - LLC Medical Technologies, Saint Petersburg
  - St. Petersburg State Pediatric Medical University, Saint Petersburg
  - "Baltiyskaya Medicyna" LLC, Saint Petersburg
  - RSBHI Smolensk Regional Clinical Hospital, Smolensk
  - SHI Ulyanovsk Regional Children's Clinical Hospital n. a. Y.F.Goryachev, Ulyanovsk
  - SHI Central Clinical Medical Unit, Ulyanovsk
  - MAI Children's City Clinical Hospital 9, Yekaterinburg
- Serbia (3):
  - Institute for Child and Youth Healthcare of Vojvodina, Novi Sad, Vojvodina
  - Mother and Child Healthcare Institute Dr Vukan Cupic, Belgrade
  - University Children's Hospital Belgrade, Belgrade
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Hospital Universitario Miguel Servet, Zaragoza, Spain
- Taiwan (3):
  - Chang Gung Memorial Hospital- Kaohsiung branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Thailand (2):
  - Siriraj Hospital, Faculty of Medicine, Mahidol University, Bangkoknoi, Bangkok
  - Phramongkutklao Hospital, Ratchathevee, Bangkok
- Turkey (Türkiye) (3):
  - Izmir Tepecik Training and Research Hospital, Izmir, Konak
  - Eskisehir Osmangazi Universitesi Tip Fakultesi, Eskişehir
  - Karadeniz Teknik Universitesi Tip Fakultesi Farabi Hastanesi, Trabzon
- Ukraine (5):
  - Komunalnyi zaklad "Dnipropetrovska dytiacha miska klinichna likarnia #5", Dnipro
  - Komunalnyi zaklad "Dnipropetrovska oblasna dytiacha klinichna likarnia", Dnipro
  - Ivano-Frankivska oblasna dytiacha klinichna likarnia, Ivano-Frankivsk
  - DZ "Ukrainskyi medychnyi tsentr reabilitatsii ditei z orhanichnym urazhenniam, Kyiv
  - Oblasnyi klinichnyi tsentr neirokhirurhii ta nevrolohii,viddilennia neirokhirurhii #2, Uzhhorod

REFERENCES:
- [Derived] Mann D, Antinew J, Knapp L, Almas M, Liu J, Scavone J, Yang R, Modequillo M, Makedonska I, Ortiz M, Kyrychenko A, Nordli D, Farkas V, Farkas MK; A0081042 study group. Pregabalin adjunctive therapy for focal onset seizures in children 1 month to <4 years of age: A double-blind, placebo-controlled, video-electroencephalographic trial. Epilepsia. 2020 Apr;61(4):617-626. doi: 10.1111/epi.16466. Epub 2020 Mar 18. PMID 32189338
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081042&StudyName=A%20Safety%2C%20Efficacy%2C%20and%20Tolerability%20Trial%20of%20Pregabalin%20as%20Add-On%20Treatment%20in%20Pediatric%20Subjects%20%3C4%20years%20of%20age%20with%20Partial%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received treatment in double-blind treatment phase (total duration: 21 days) which included dose escalation (5 days), fixed-dose (9 days) and taper (7 days).
Groups:
- Pregabalin 7 mg/kg/Day or 6 mg/kg/Day: Participants aged greater than (>) 3 months to less than (<) 4 years, received Pregabalin 3.5 milligrams per kilogram per day (mg/kg/day) (3.0 mg/kg/day for participants 1 to 3 months of age), orally three times daily (TID) in equally divided doses for first 5 days; followed by 7 mg/kg/day (6 mg/kg/day for participants 1 to 3 months of age), orally TID in equally divided doses for 9 days and 3.5 mg/kg/day (3.0 mg/kg/day for participants 1 to 3 months of age), orally TID in equally divided doses for next 7 days.
- Pregabalin 14 mg/kg/Day or 12 mg/kg/Day: Participants aged >3 months to <4 years, received Pregabalin 3.5 mg/kg/day (3.0 mg/kg/day for participants 1 to 3 months of age), orally TID in equally divided doses for first 2 days and 7 mg/kg/day (6 mg/kg/day for participants 1 to 3 months of age), orally TID in equally divided doses for next 3 days; followed by 14 mg/kg/day (12 mg/kg/day for participants 1 to 3 months of age), orally TID in equally divided doses for 9 days; and 7 mg/kg/day (6 mg/kg/day for participants 1 to 3 months of age), orally TID in equally divided doses for next 4 days and 3.5 mg/kg/day (3.0 mg/kg/day for participants 1 to 3 months of age), orally TID in equally divided doses for next 3 days.
- Placebo: Participants aged >3 months to <4 years received placebo matched to Pregabalin, orally TID for 21 days.
Period: Overall Study
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Started | 71 | 34 | 70
Completed | 69 | 33 | 67
Not Completed | 2 | 1 | 3
Not completed — Insufficient clinical response | 1 | 0 | 1
Not completed — No longer willing to participate | 1 | 0 | 1
Not completed — Medication error | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Pregabalin 7 mg/kg/Day or 6 mg/kg/Day: Participants aged > 3 months to < 4 years, received Pregabalin 3.5 mg/kg/day (3.0 mg/kg/day for participants 1 to 3 months of age), orally TID in equally divided doses for first 5 days; followed by 7 mg/kg/day (6 mg/kg/day for participants 1 to 3 months of age), orally TID in equally divided doses for 9 days and 3.5 mg/kg/day (3.0 mg/kg/day for participants 1 to 3 months of age), orally TID in equally divided doses for next 7 days.
- Total: Total of all reporting groups
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo | Total
Number analyzed (Participants) | 71 | 34 | 70 | 175
Age, Continuous [Mean (Standard Deviation); unit: months] | 27.5 (12.7) | 28.5 (12.5) | 28.8 (12.6) | 28.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 14 | 32 | 72
  Male | 45 | 20 | 38 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 23 | 10 | 19 | 52
  White | 47 | 24 | 49 | 120
  Other | 1 | 0 | 2 | 3
Weight [Mean (Standard Deviation); unit: kilogram] | 11.7 (3.5) | 11.4 (3.4) | 11.4 (3.1) | 11.5 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Log Transformed 24-Hour Seizure Rate for All Partial Onset Seizures During the Double-Blind Treatment Phase
Description: All partial onset seizures experienced during treatment phase were recorded by central reader during the 48 to 72 hour video-electroencephalogram (EEG). Double Blind 24 hour EEG seizure rate for all partial onset seizures = ([Number of seizures in double blind 48 to 72 hour EEG assessment] divided by [number of hours of video-EEG monitoring])*24. The EEG assessment was done at the end of the fixed dose treatment. For log-transformation, the quantity 1 was added to the double blind 24 hour EEG seizure rate for all participants to account for any possible "0" seizure incidence. This resulted in final calculation as: log transformed (double-blind 24-hour EEG seizure rate + 1).
Time Frame: Day 1 up to Day 14
Population: Modified intent-to-treat (mITT) population included all randomized participants who took at least one dose of study drug during the double-blind treatment phase, had a baseline with at least one partial onset seizure identified by video-EEG (at least 24 hours of evaluable monitoring) and a treatment phase video-EEG.
Measure: Least Squares Mean (Standard Error); unit: seizures per 24 hours
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Number analyzed (Participants) | 59 | 28 | 53
seizures per 24 hours | 1.69 (0.115) | 1.15 (0.163) | 1.58 (0.129)
Statistical Analysis 1: Comparison: Pregabalin 7 mg/kg/Day or 6 mg/kg/Day vs Placebo; Linear model with log transformed baseline seizure rate as continuous covariate and treatment, age stratum, and geographical region as fixed factor effects; Test type: Superiority; p = 0.4606, ANCOVA; Least Square Mean Difference = 0.11, 95% CI 2-sided [-0.19 to 0.42], Standard Error of Mean 0.153
Statistical Analysis 2: Comparison: Pregabalin 14 mg/kg/Day or 12 mg/kg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0223, ANCOVA; Least Square Mean Difference = -0.43, 95% CI 2-sided [-0.80 to -0.06], Standard Error of Mean 0.185

2. Secondary Outcome: Responder Rate: Percentage of Participants With at Least 50 Percent (%) or Greater Reduction From Baseline in 24-Hour Seizure Rate for All Partial Onset Seizures During the Double-Blind Treatment Phase
Description: Responder Rate was defined as percentage of participants who had a 50% or greater reduction from baseline in 24-hour seizure rate during the double-blind treatment phase. Double Blind 24 hour EEG seizure rate for all partial onset seizures = ([Number of seizures in double blind 48 to 72 hour EEG assessment] divided by [number of hours of video-EEG monitoring])*24. The EEG assessment was done at the end of the fixed dose treatment.
Time Frame: Day 1 up to Day 14
Population: mITT population included all randomized participants who took at least one dose of study drug during the double-blind treatment phase, had a baseline with at least one partial onset seizure identified by Video-EEG (at least 24 hours of evaluable monitoring) and a treatment phase Video-EEG.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Number analyzed (Participants) | 59 | 28 | 53
percentage of participants | 30.51 | 53.57 | 41.51
Statistical Analysis 1: Comparison: Pregabalin 7 mg/kg/Day or 6 mg/kg/Day vs Placebo; The dichotomized responder variable was analyzed using a logistic regression model via maximum likelihood estimation with treatment group, age stratum, and geographical region as a fixed effect covariates; Test type: Superiority; p = 0.2418, Regression, Logistic; Odds Ratio (OR) = 0.625, 95% CI 2-sided [0.284 to 1.373]
Statistical Analysis 2: Comparison: Pregabalin 14 mg/kg/Day or 12 mg/kg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3050, Regression, Logistic; Odds Ratio (OR) = 1.622, 95% CI 2-sided [0.644 to 4.086]

3. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were events which occurred between first dose of study drug and up to end of study (up to Day 25) that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Day 1 up to End of study (EOS) (maximum Day 25)
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Number analyzed (Participants) | 71 | 34 | 70
Participants
  AEs | 32 | 17 | 38
  SAEs | 0 | 1 | 4

4. Other Pre Specified Outcome: Number of Participants With Treatment-Related Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were events which occurred between first dose of study drug and up to end of study (up to Day 25) that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to drug was assessed by the investigator. AEs included both serious and non-serious adverse events.
Time Frame: Day 1 up to EOS (maximum Day 25)
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Number analyzed (Participants) | 71 | 34 | 70
Participants
  AEs | 15 | 8 | 13
  SAEs | 0 | 0 | 1

5. Other Pre Specified Outcome: Number of Adverse Events by Severity
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs were classified according to the severity in 3 categories a) mild: AEs does not interfere with participant's usual function b) moderate: AEs interferes to some extent with participant's usual function c) severe: AEs interferes significantly with participant's usual function.
Time Frame: Day 1 up to EOS (maximum Day 25)
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: events
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Number analyzed (Participants) | 71 | 34 | 70
events
  Mild | 60 | 23 | 67
  Moderate | 3 | 13 | 19
  Severe | 0 | 0 | 0

6. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Abnormality Criteria: hemoglobin,hematocrit,red blood cells(RBC)count:<0.8*lower limit of normal[LLN],platelets:<0.5*LLN/>1.75*upper limit of normal[ULN]; leukocytes:<0.6*LLN/>1.5*ULN; lymphocytes,neutrophils, total protein,albumin, tetraiodothyronine,thyroid stimulating hormone:<0.8*LLN/>1.2*ULN; basophils,eosinophils,monocytes:>1.2*ULN; prothrombin [PT],PT international ratio:>1.1*ULN; aspartate aminotransferase,alanine aminotransferase,alkaline phosphatase,gamma glutamyl transferase:>0.3*ULN; bilirubin:>1.5*ULN; blood urea nitrogen,creatinine, cholesterol,triglycerides:>1.3*ULN; sodium: <0.95*LLN/>1.05*ULN; potassium,chloride,calcium,bicarbonate:<0.9*LLN/>1.1*ULN; glucose fasting:<0.6*LLN/>1.5*ULN; creatine kinase:>2*ULN;urine glucose,ketone,protein:>=1;urine WBC,RBC:>= 20/High Power Field[HPF]; urine casts,hyaline casts:>1/Low Power Field; urine bacteria:>20/HPF.
Time Frame: From Baseline up to EOS (maximum Day 25)
Population: Safety population included all randomized participants who received at least 1 dose of study drug. Here, "Overall number of participants analyzed"= number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Number analyzed (Participants) | 71 | 34 | 69
Participants | 65 | 29 | 61

7. Other Pre Specified Outcome: Number of Participants With Vital Signs Abnormalities
Description: Criteria for abnormalities in vital signs included: sitting/supine systolic blood pressure (SBP) values: maximum increase and decrease of greater than or equal to (>=) 30 millimeter of mercury (mmHg) from baseline; sitting/supine diastolic blood pressure (DBP) value: maximum increase and decrease of >=20 mmHg from baseline.
Time Frame: From Baseline (BL) up to EOS (maximum Day 25)
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Number analyzed (Participants) | 71 | 34 | 70
Participants
  Maximum Increase from BL(>=30):sitting/supine SBP | 2 | 0 | 1
  Maximum Increase from BL(>=20):sitting/supine DBP | 7 | 1 | 3
  Maximum Decrease from BL(>=30):sitting/supine SBP | 1 | 0 | 1
  Maximum Decrease from BL(>=20):sitting/supine DBP | 2 | 2 | 1

8. Other Pre Specified Outcome: Percentage of Participants With Abnormal Physical Examination Findings at Screening and End of Study
Description: Physical examinations evaluated the following body systems/organs: abdomen; ears; extremities; eyes; general appearance; head; heart; lungs; lymph nodes; mouth; musculoskeletal; nose; skin and throat. Abnormalities in physical examination were based on investigator's discretion.
Time Frame: Screening and EOS (maximum Day 25)
Population: Safety population included all randomized participants who received at least 1 dose of study drug. Here, "number analyzed" signifies number of participants who were evaluable for the specified category for each arm respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Number analyzed (Participants) | 71 | 34 | 70
percentage of participants
  Abdomen: Screening | 4.2 | 5.9 | 2.9
  Abdomen: EOS: number analyzed (Participants) | 71 | 34 | 69
  Abdomen: EOS | 4.2 | 5.9 | 1.4
  Ears: Screening | 1.4 | 0 | 1.4
  Ears: EOS: number analyzed (Participants) | 70 | 34 | 69
  Ears: EOS | 1.4 | 0 | 1.4
  Extremities: Screening | 14.1 | 26.5 | 15.7
  Extremities: EOS: number analyzed (Participants) | 71 | 34 | 69
  Extremities: EOS | 14.1 | 26.5 | 18.8
  Eyes: Screening | 9.9 | 20.6 | 17.1
  Eyes: EOS: number analyzed (Participants) | 71 | 34 | 69
  Eyes: EOS | 9.9 | 20.6 | 18.8
  General appearance: Screening | 15.5 | 26.5 | 15.7
  General appearance: EOS: number analyzed (Participants) | 71 | 34 | 69
  General appearance: EOS | 15.5 | 23.5 | 15.9
  Head: Screening | 31.0 | 47.1 | 31.4
  Head: EOS: number analyzed (Participants) | 71 | 34 | 69
  Head: EOS | 33.8 | 47.1 | 31.9
  Heart: Screening | 1.4 | 8.8 | 4.3
  Heart: EOS: number analyzed (Participants) | 71 | 34 | 69
  Heart: EOS | 1.4 | 5.9 | 4.3
  Lungs: Screening | 2.8 | 8.8 | 4.3
  Lungs: EOS: number analyzed (Participants) | 71 | 34 | 69
  Lungs: EOS | 2.8 | 8.8 | 5.8
  Lymph nodes: Screening | 0 | 8.8 | 0
  Lymph nodes: EOS: number analyzed (Participants) | 70 | 34 | 69
  Lymph nodes: EOS | 0 | 2.9 | 0
  Mouth: Screening | 9.9 | 2.9 | 5.7
  Mouth: EOS: number analyzed (Participants) | 70 | 34 | 69
  Mouth: EOS | 7.1 | 2.9 | 5.8
  Musculoskeletal: Screening | 31.0 | 38.2 | 35.7
  Musculoskeletal: EOS: number analyzed (Participants) | 71 | 34 | 69
  Musculoskeletal: EOS | 33.8 | 38.2 | 37.7
  Nose: Screening | 0 | 2.9 | 0
  Nose: EOS: number analyzed (Participants) | 70 | 34 | 69
  Nose: EOS | 0 | 0 | 5.8
  Skin: Screening | 9.9 | 14.7 | 21.4
  Skin: EOS: number analyzed (Participants) | 71 | 34 | 69
  Skin: EOS | 8.5 | 14.7 | 21.7
  Throat: Screening | 1.4 | 2.9 | 0
  Throat: EOS: number analyzed (Participants) | 70 | 34 | 68
  Throat: EOS | 0 | 5.9 | 2.9

9. Other Pre Specified Outcome: Percentage of Participants With Abnormal Neurological Examination Findings at Baseline and End of Study
Description: Neurological examinations included: coordination; cranial nerve function (CNF); gait and station; level of consciousness (LOC); lower and upper extremity sensation; muscle strength; muscle tone; nystagmus; reflexes and speech. Abnormalities in neurological examination were based on investigator's discretion and also, some components of the neurological examination were not done for certain participants due to participant age or significant developmental impairment. Only those categories of neurological examination in which at least 10% of participants had an abnormality in any treatment group at any time point were reported in this outcome measure.
Time Frame: Baseline (BL) and EOS (maximum Day 25)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Number analyzed (Participants) | 71 | 34 | 70
percentage of participants
  Coordination- left hand movement (BL) | 1.4 | 11.8 | 8.6
  Coordination-left hand movement (EOS): number analyzed (Participants) | 71 | 34 | 69
  Coordination-left hand movement (EOS) | 1.4 | 8.8 | 10.1
  Coordination- right hand movement (EOS): number analyzed (Participants) | 71 | 34 | 69
  Coordination- right hand movement (EOS) | 2.8 | 5.9 | 10.1
  Coordination- romberg test (BL) | 2.8 | 8.8 | 10.0
  Coordination- romberg test (EOS): number analyzed (Participants) | 71 | 34 | 69
  Coordination- romberg test (EOS) | 2.8 | 5.9 | 11.6
  CNF- left eye visual field (BL) | 12.7 | 8.8 | 10.0
  CNF- left eye visual field (EOS): number analyzed (Participants) | 71 | 34 | 69
  CNF- left eye visual field (EOS) | 12.7 | 8.8 | 10.1
  CNF: right eye visual field (BL) | 12.7 | 5.9 | 10.0
  CNF: right eye visual field (EOS): number analyzed (Participants) | 71 | 34 | 69
  CNF: right eye visual field (EOS) | 12.7 | 5.9 | 10.1
  CNF: left fundoscopic exam (BL) | 12.7 | 26.5 | 12.9
  CNF: left fundoscopic exam (EOS): number analyzed (Participants) | 71 | 34 | 69
  CNF: left fundoscopic exam (EOS) | 12.7 | 23.5 | 14.5
  CNF: right fundoscopic exam (BL) | 11.3 | 20.6 | 14.3
  CNF: right fundoscopic exam (EOS): number analyzed (Participants) | 71 | 34 | 69
  CNF: right fundoscopic exam (EOS) | 11.3 | 17.6 | 14.5
  CNF: left visual acuity (BL) | 11.3 | 11.8 | 12.9
  CNF: left visual acuity (EOS): number analyzed (Participants) | 71 | 34 | 69
  CNF: left visual acuity (EOS) | 11.3 | 11.8 | 13.0
  CNF: right visual acuity (BL) | 11.3 | 11.8 | 11.4
  CNF: right visual acuity (EOS): number analyzed (Participants) | 71 | 34 | 69
  CNF: right visual acuity (EOS) | 11.3 | 11.8 | 11.6
  CNF: finger tracking (BL) | 22.5 | 26.5 | 24.3
  CNF: finger tracking (EOS): number analyzed (Participants) | 71 | 34 | 69
  CNF: finger tracking (EOS) | 21.1 | 23.5 | 26.1
  CNF: swallowing (BL) | 14.1 | 14.7 | 14.3
  CNF: swallowing (EOS): number analyzed (Participants) | 71 | 34 | 69
  CNF: swallowing (EOS) | 14.1 | 14.7 | 14.5
  CNF:Left shoulder,head turn strength (BL) | 11.3 | 2.9 | 7.1
  CNF: Left shoulder shrug,head turn strength (EOS): number analyzed (Participants) | 71 | 34 | 69
  CNF: Left shoulder shrug,head turn strength (EOS) | 11.3 | 2.9 | 10.1
  Gait and station - gait (BL) | 52.1 | 50.0 | 45.7
  Gait and station - gait (EOS): number analyzed (Participants) | 71 | 34 | 69
  Gait and station - gait (EOS) | 52.1 | 52.9 | 46.4
  Level of consciousness (BL) | 5.6 | 20.6 | 5.7
  Level of consciousness (EOS): number analyzed (Participants) | 71 | 34 | 69
  Level of consciousness (EOS) | 7.0 | 20.6 | 2.9
  Muscle strength -lower extremities (BL) | 49.3 | 58.8 | 51.4
  Muscle strength -lower extremities (EOS): number analyzed (Participants) | 71 | 34 | 69
  Muscle strength -lower extremities (EOS) | 49.3 | 58.8 | 53.6
  Muscle strength - upper extremities (BL) | 47.9 | 58.8 | 50.0
  Muscle strength - upper extremities (EOS): number analyzed (Participants) | 71 | 34 | 69
  Muscle strength - upper extremities (EOS) | 49.3 | 58.8 | 52.2
  Muscle strength - trunk (BL) | 43.7 | 38.2 | 44.3
  Muscle strength - trunk (EOS): number analyzed (Participants) | 71 | 34 | 69
  Muscle strength - trunk (EOS) | 39.4 | 38.2 | 42.0
  Muscle tone - lower extremities (BL): number analyzed (Participants) | 70 | 34 | 69
  Muscle tone - lower extremities (BL) | 64.3 | 73.5 | 63.8
  Muscle tone - lower extremities (EOS): number analyzed (Participants) | 71 | 34 | 68
  Muscle tone - lower extremities (EOS) | 64.8 | 73.5 | 66.2
  Muscle tone - upper extremities (BL): number analyzed (Participants) | 71 | 34 | 69
  Muscle tone - upper extremities (BL) | 64.8 | 73.5 | 63.8
  Muscle tone - upper extremities (EOS): number analyzed (Participants) | 71 | 34 | 68
  Muscle tone - upper extremities (EOS) | 64.8 | 73.5 | 66.2
  Nystagmus - horizontal (BL) | 9.9 | 11.8 | 7.1
  Nystagmus - horizontal (EOS): number analyzed (Participants) | 71 | 34 | 69
  Nystagmus - horizontal (EOS) | 8.5 | 11.8 | 5.8
  Reflexes - left ankle (BL) | 46.5 | 52.9 | 47.1
  Reflexes - left ankle (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - left ankle (EOS) | 46.5 | 52.9 | 46.4
  Reflexes - right ankle (BL) | 46.5 | 58.8 | 47.1
  Reflexes - right ankle (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - right ankle (EOS) | 45.1 | 58.8 | 46.4
  Reflexes - left babinski (BL) | 42.3 | 47.1 | 47.1
  Reflexes - left babinski (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - left babinski (EOS) | 40.8 | 47.1 | 47.8
  Reflexes - right babinski (BL) | 42.3 | 55.9 | 50.0
  Reflexes - right babinski (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - right babinski (EOS) | 40.8 | 55.9 | 50.7
  Reflexes - left biceps (BL) | 47.9 | 52.9 | 50.0
  Reflexes - left biceps (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - left biceps (EOS) | 47.9 | 52.9 | 49.3
  Reflexes - right biceps (BL) | 46.5 | 58.8 | 52.9
  Reflexes - right biceps (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - right biceps (EOS) | 46.5 | 58.8 | 52.2
  Reflexes - left brachioradialis (BL) | 45.1 | 52.9 | 48.6
  Reflexes - left brachioradialis (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - left brachioradialis (EOS) | 45.1 | 52.9 | 47.8
  Reflexes - right brachioradialis (BL) | 43.7 | 58.8 | 50.0
  Reflexes - right brachioradialis (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - right brachioradialis (EOS) | 43.7 | 58.8 | 50.7
  Reflexes - left knee (BL) | 53.5 | 55.9 | 57.1
  Reflexes - left knee (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - left knee (EOS) | 52.1 | 58.8 | 56.5
  Reflexes - right knee (BL) | 52.1 | 61.8 | 61.4
  Reflexes - right knee (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - right knee (EOS) | 50.7 | 64.7 | 59.4
  Reflexes - left triceps (BL) | 46.5 | 52.9 | 45.7
  Reflexes - left triceps (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - left triceps (EOS) | 46.5 | 52.9 | 44.9
  Reflexes - right triceps (BL) | 45.1 | 58.8 | 48.6
  Reflexes - right triceps (EOS): number analyzed (Participants) | 71 | 34 | 69
  Reflexes - right triceps (EOS) | 45.1 | 58.8 | 47.8
  Speech - articulation (BL) | 53.5 | 47.1 | 45.7
  Speech - articulation (EOS): number analyzed (Participants) | 71 | 34 | 69
  Speech - articulation (EOS) | 54.9 | 44.1 | 47.8
  Speech - language (BL) | 69.0 | 76.5 | 65.7
  Speech - language (EOS): number analyzed (Participants) | 71 | 34 | 69
  Speech - language (EOS) | 69.0 | 73.5 | 66.7

10. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for abnormalities in ECG findings: 1) Time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS complex): >=140 milliseconds (msec); 2) The interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization (PR interval): >=200 msec; 3) Time from ECG Q wave to the end of the T wave corresponding to electrical systole corrected for heart rate using Fridericia's formula (QTCF interval): absolute value 450 to <480 msec, 480 to <500 msec, >=500 msec; 4) Maximum QT interval: >=500 msec; 5) Maximum QTCB interval (Bazett's correction): 450 to< 480 msec, 480 to <500 msec, >=500 msec. Only those categories of ECG abnormalities in which participants were found abnormal (maximum QTCB interval 450-<480 msec), were reported in this outcome measure.
Time Frame: From screening up to EOS (maximum Day 25)
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
Number analyzed (Participants) | 71 | 34 | 70
Participants | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to End of Study (maximum Day 25)
Arm/Group | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/34 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/71 | 1/34 | 4/70
Other Adverse Events (participants affected / at risk) | 32/71 | 16/34 | 37/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day (N=71) | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day (N=34) | Placebo (N=70)
Pneumonia (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 7 mg/kg/Day or 6 mg/kg/Day (N=71) | Pregabalin 14 mg/kg/Day or 12 mg/kg/Day (N=34) | Placebo (N=70)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Chalazion (Eye disorders) | 1 | 0 | 0
Mydriasis (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Oral contusion (Gastrointestinal disorders) | 1 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 6
Application site irritation (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Hyperthermia (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 2 | 4
Sluggishness (General disorders) | 0 | 0 | 1
Feeling hot (General disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Bronchitis viral (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 1 | 0 | 0
Lice infestation (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 3
Otitis media (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Respiratory tract infection viral (Infections and infestations) | 2 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 8
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Viral infection (Infections and infestations) | 2 | 2 | 2
Viral rash (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Lymphocyte morphology abnormal (Investigations) | 1 | 0 | 0
Lymphocyte percentage increased (Investigations) | 1 | 0 | 0
Neutrophil percentage decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0
Myoclonic epilepsy (Nervous system disorders) | 0 | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 2 | 3
Somnolence (Nervous system disorders) | 8 | 6 | 4
Agitation (Psychiatric disorders) | 0 | 0 | 1
Enuresis (Psychiatric disorders) | 0 | 0 | 1
Irritability (Psychiatric disorders) | 3 | 0 | 1
Sleep disorder (Psychiatric disorders) | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT02072824/SAP_000.pdf
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT02072824/Prot_001.pdf